CLINICAL TRIAL: NCT00434122
Title: A Randomised, Assessor-blind, Parallel Groups, Multi-centre, Exploratory Study Assessing the Impact of Subcutaneous Administration of Degarelix 2.5 mg on Synchronisation of Follicle Cohort Compared to Placebo and Evaluating the Effects of Degarelix 2.5 mg Started in the Mid-luteal or Early Follicular Phase on Endometrial Receptivity Compared to a Fixed Gonadotrophin Releasing Hormone Antagonist Protocol in Oocyte Donors Undergoing Controlled Ovarian Hyperstimulation for Assisted Reproductive Technologies
Brief Title: Exploratory Study Assessing Synchronisation of Egg Sacs With Degarelix
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FE200486 CS24
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Results first posted 2009-04-10 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Infertility, Female
Keywords: Assisted Reproductive Technology (ART); oocyte donors undergoing controlled ovarian hyperstimulation for assisted reproductive technologies
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Degarelix mid-luteal, 2.5 mg (Experimental): Degarelix 2.5 mg will be injected subcutaneously (SC) 7 days after luteinizing hormone (LH) peak and on Stimulation Day 6. Placebo will be injected SC on Stimulation Day 1.
  Interventions: Drug: Degarelix mid-luteal, 2.5 mg
- Placebo (Placebo Comparator): Placebo will be injected subcutaneously (SC) 7 days after luteinizing hormone (LH) peak. Degarelix 2.5 mg will be injected SC on Stimulation Day 1 and Stimulation Day 6.
  or Placebo will be injected SC 7 days after LH peak and on Stimulation Day 1. Ganirelix 0.25 mg will be injected SC daily from Stimulation Day 6 until the last stimulation day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Degarelix mid-luteal, 2.5 mg — Degarelix 2.5 mg will be injected subcutaneously (SC) 7 days after luteinizing hormone (LH) peak and on Stimulation Day 6. Placebo will be injected SC on Stimulation Day 1.
  Arms: Degarelix mid-luteal, 2.5 mg
Drug: Placebo — Placebo will be injected subcutaneously (SC) 7 days after luteinizing hormone (LH) peak. Degarelix 2.5 mg will be injected SC on Stimulation Day 1 and Stimulation Day 6.
  or Placebo will be injected SC 7 days after LH peak and on Stimulation Day 1. Ganirelix 0.25 mg will be injected SC daily from Stimulation Day 6 until the last stimulation day.
  Arms: Placebo

SUMMARY:
The main purpose of this clinical research study is to investigate if degarelix can synchronise the growth of the egg sacs in the ovaries and if degarelix has any effect on the lining of the womb.

DETAILED DESCRIPTION:
For the primary end-point (data collected on Stimulation Day 1), the study will compare degarelix 2.5 mg administered in the mid-luteal phase to placebo administered in the mid-luteal phase.

After Stimulation Day 1 the placebo group will be split into two groups: a degarelix 2.5 mg follicular group and a ganirelix 0.25 mg group.

ELIGIBILITY:
Inclusion Criteria

* Signed Informed Consent Form, prior to screening evaluations
* In good physical and mental health
* Pre-menopausal females between the ages of 18-35 years (both inclusive) at the time of randomisation
* Regular menstrual cycles of 26-35 days duration (both inclusive), presumed to be ovulatory
* Body mass index (BMI) between 18 and 29 kg/m2 (both inclusive)
* Willing to donate the retrieved oocytes
* Willing to use an adequate barrier method of contraception from informed consent to Day hCG injection +7 and to use an adequate barrier or hormonal method of contraception from Day hCG injection +7 to the end-of-study visit

Exclusion Criteria

* Abnormal karyotype
* Any known clinically significant systemic disease (e.g., insulin dependent diabetes)
* Any known endocrine or metabolic abnormalities (pituitary, adrenal, pancreas, liver or kidney) which can compromise participation in the study
* Diagnosed with polycystic ovarian syndrome or endometriosis stage III/IV
* Diagnosed as "poor responder"
* History of recurrent miscarriage (defined as three consecutive spontaneous losses before weeks 24 of pregnancy)
* Pregnancy or lactation
* Use of any investigational drug during 3 months prior to start of the current COH cycle
* Previous participation in the study
* Hypersensitivity to any trial product

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (4):
- UZ Brussel, Brussels, Belgium
- ISCARE IVF a.s., Prague, Czechia
- Spain (2):
  - IVI-Madrid, Madrid
  - IVI-Valencia, Valencia

REFERENCES:
- [Derived] Garcia-Velasco JA, Kupesic S, Pellicer A, Bourgain C, Simon C, Mrazek M, Devroey P, Arce JC. Follicular and endocrine profiles associated with different GnRH-antagonist regimens: a randomized controlled trial. Reprod Biomed Online. 2012 Feb;24(2):153-62. doi: 10.1016/j.rbmo.2011.10.016. Epub 2011 Nov 4. PMID 22197127

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Degarelix Mid-luteal, 2.5 mg | Placebo
Started | 42 (Randomised) | 43 (Randomised)
Intention-to-treat (ITT) Population | 39 (All randomised and exposed subjects not withdrawn before Stimulation Day 1.) | 39 (All randomised and exposed subjects not withdrawn before Stimulation Day 1.)
Completed | 36 | 36
Not Completed | 6 | 7
Not completed — Non-compliance with protocol | 0 | 1
Not completed — loss of subject contact | 1 | 1
Not completed — Personal reasons | 1 | 1
Not completed — Large follicle size | 2 | 2
Not completed — Low follicular response. | 1 | 2
Not completed — Travelling of subject. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix Mid-luteal, 2.5 mg | Placebo | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Categorical [Count of Participants; unit: Participants] — Intention-to-treat (ITT) population
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 39 | 39 | 78
    >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] — ITT population
  years | 28.9 (4.1) | 28.0 (3.9) | 28.4 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants] — ITT population
  Participants
    Female | 39 | 39 | 78
    Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — ITT population
  participants
    Czech Republic | 7 | 7 | 14
    Spain | 27 | 26 | 53
    Belgium | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Coefficient of Variation of Follicular Sizes on Stimulation Day 1 (Follicles ≥ 2 mm)
Description: Explanation of the term "coefficient of variation": The coefficient of variation is a normalized measure of dispersion of a probability distribution.
Time Frame: Stimulation Day 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Degarelix Mid-luteal, 2.5 mg | Placebo
Number analyzed (Participants) | 39 | 39
Percentage | 36.7 (5.6) | 39.2 (9.5)

2. Secondary Outcome: Frequency of Oocyte Donors With Adequate Secretory Transformation at the Endometrial Histology Evaluation 7 Days After Injection With Human Chorionic Gonadotrophin (hCG)
Description: An adequate secretory endometrium 7 days after hCG injection was defined as secretory in the histological classification and with endometrial dating corresponding to the expected cycle day ±1 day.
Time Frame: 7 days after hCG injection
Population: Subjects with evaluable endometrial biopsies 7 days after injection with hCG.
Measure: Number; unit: Participants
Groups:
- Degarelix Follicular, 2.5 mg: Placebo will be injected subcutaneously (SC) 7 days after luteinizing hormone (LH) peak. Degarelix 2.5 mg will be injected SC on Stimulation Day 1 and Stimulation Day 6
- Ganirelix, 0.25 mg: Placebo will be injected subcutaneously (SC) 7 days after luteinizing hormone (LH) peak and on Stimulation Day 1. Ganirelix 0.25 mg will be injected SC daily from Stimulation Day 6 until the last stimulation day.
Arm/Group | Degarelix Mid-luteal, 2.5 mg | Degarelix Follicular, 2.5 mg | Ganirelix, 0.25 mg
Number analyzed (Participants) | 32 | 14 | 16
Participants | 31 | 11 | 14

ADVERSE EVENTS:
Time Frame: From signed informed consent till end-of-trial visit (approximately 12 +/- 2 weeks after oocyte retrieval)
Description: Evaluated at each trial visit
Groups:
- Degarelix, 2.5 mg: Combination of these two groups: Degarelix Mid-luteal 2.5 mg and Degarelix Follicular 2.5 mg.
  Degarelix Mid-luteal, 2.5 mg: Degarelix 2.5 mg will be injected subcutaneously (SC) 7 days after luteinizing hormone (LH) peak and on Stimulation Day 6. Placebo will be injected SC on Stimulation Day 1.
  Degarelix Follicular, 2.5 mg: Placebo will be injected subcutaneously (SC) 7 days after luteinizing hormone (LH) peak. Degarelix 2.5 mg will be injected SC on Stimulation Day 1 and Stimulation Day 6.
- Ganirelix, 0.25 mg: Placebo will be injected SC 7 days after LH peak and on Stimulation Day 1. Ganirelix 0.25 mg will be injected SC daily from Stimulation Day 6 until the last stimulation day.
Arm/Group | Degarelix, 2.5 mg | Ganirelix, 0.25 mg
Serious Adverse Events (participants affected / at risk) | 1/63 | 0/22
Other Adverse Events (participants affected / at risk) | 7/63 | 4/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix, 2.5 mg (N=63) | Ganirelix, 0.25 mg (N=22)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix, 2.5 mg (N=63) | Ganirelix, 0.25 mg (N=22)
Injection site erythema (General disorders) | 3 (3) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 3 (3) | 0 (0)
Menstruation delayed (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restiction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.